CLINICAL TRIAL: NCT00236119
Title: A 12-Week, Exploratory, Open-Label, Nonrandomized, Dose-Escalation Study of the Efficacy, Safety and Tolerability of Oral CEP-701 in Patients With Severe, Recalcitrant, Plaque Type Psoriasis
Brief Title: Study of the Efficacy, Safety and Tolerability of Oral CEP-701 in Patients With Severe Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cephalon (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: C0701/2024/DR/US
Record Dates: First submitted 2005-10-11; First posted 2005-10-12 (Estimated); Last update posted 2012-08-23 (Estimated); Status verified 2012-08

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — lestaurtinib

ARMS (4):
- CEP-701 20mg (Experimental): Patient Cohort 1
  Interventions: Drug: CEP-701 20mg
- CEP-701 40mg (Experimental): Patient Cohort 2
  Interventions: Drug: CEP-701 20mg; Drug: CEP-701 40mg
- CEP-701 60mg (Experimental): Patient Cohort 3
  Interventions: Drug: CEP-701 20mg; Drug: CEP-701 40mg; Drug: CEP-701 60mg
- CEP-701 80mg (Experimental): Patient Cohort 4
  Interventions: Drug: CEP-701 20mg; Drug: CEP-701 40mg; Drug: CEP-701 60mg; Drug: CEP-701 80mg

INTERVENTIONS:
Drug: CEP-701 20mg — Dosages of oral CEP-701 20mg will be given twice daily. Escalation to the next higher dosage, CEP-701 40mg, may occur once the first 8 patients at the current dosage have completed 8 weeks of treatment without adverse events or laboratory abnormalities. Patients who remain in Cohort 1 will continue on the 20mg dosage until study completion.
Drug: CEP-701 40mg — Dosages of oral CEP-701 40mg will be given twice daily.Escalation to the next higher dosage, CEP-701 60mg, may occur once 8 weeks of treatment at the current dosage is completed without adverse events or laboratory abnormalities. Patients who remain in Cohort 2 will continue on the 40mg dosage until study completion.
  Arms: CEP-701 40mg; CEP-701 60mg; CEP-701 80mg
Drug: CEP-701 60mg — Dosages of oral CEP-701 60mg will be given twice daily. Escalation to the next higher dosage, CEP-701 80mg, may occur once 8 weeks of treatment at the current dosage is completed without adverse events or laboratory abnormalities. Patients who remain in Cohort 3 will continue on the 60mg dosage until study completion.
  Arms: CEP-701 60mg; CEP-701 80mg
Drug: CEP-701 80mg — Dosages of oral CEP-701 80mg will be given twice daily. Patients who have moved to Cohort 4 will continue on the 80mg dosage until study completion.
  Arms: CEP-701 80mg

SUMMARY:
A 12-Week, Exploratory, Open-Label, Nonrandomized, Dose-Escalation Study of the Efficacy, Safety and Tolerability of Oral CEP-701 in Patients with Severe, Recalcitrant, Plaque Type Psoriasis.

DETAILED DESCRIPTION:
A 12-Week, Exploratory, Open-Label, Nonrandomized, Dose-Escalation Study of the Efficacy, Safety and Tolerability of Oral CEP-701 in Patients with Severe, Recalcitrant, Plaque Type Psoriasis.

ELIGIBILITY:
Inclusion Criteria:

Patients are included in the study if all of the following criteria are met:

* the patient is at least 21 years old.
* The patient has sever, recalcitrant, plaque-type psoriasis and has failed at least 1 systemic therapy (for the purposes of this study psoralen with ultraviolet light A is considered to be a systemic therapy).
* The patient has psoriatic involvement of at least 10% of BSA.
* The patient has a PSGA score of 4 or greater.
* The patient, if a woman, is surgically sterile or 2 years postmenopausal, or if of childbearing potential is currently using a medically accepted method of contraception, and agrees to continue use of this method for the duration of the study (and for 30 days after participation in the study). Acceptable methods of contraception include: abstinence, steroidal contraceptive (oral, transdermal, implanted, or injected) in conjunction with a barrier method, or intrauterine device (IUD).
* The patient, if a main, is surgically sterile, or if capable of producing offspring, is currently using an approved method of birth control, and agrees to continued use of this method for the duration of the study (and for 60 days after taking the last dose of CEP-701 because of the possible effects on spermatogenesis).
* The patient must be willing and able to comply with study procedures and restrictions and willing to return to the clinic for the follow-up evaluation as specified in this protocol.

Exclusion Criteria:

* The patient has received treatment with systemic psoriasis treatments (specifically, retinoids, methotrexate, cyclosporine A, etanercept, efalizumab, other biological agents or other immunomodulators) within 4 weeks, or UV based therapy within 2 weeks, or alefacept within 6 weeks of the planned 1st day of study treatment.
* The patient has received treatment with potent CYP3A4 inhibitors including cyclosporine, clotrimazole, fluconazole, itraconazole, ketoconazole, voriconazole, erythromycin, clarithromycin, and troleandomycin, human immunodeficiency virus (HIV) protease inhibitors, or nefazodone within 1 week (7 days) of the planned 1st day of study treatment.
* The patient is currently receiving warfarin.
* The patient has hypersensitivity to CEP-701 or any component of CEP-701.
* The patient has one or more of the following serum chemistry values as determined at the screening visit (visit 1):
* bilirubin levels greater than 2 times the upper limit of normal (ULN)
* ALT or AST levels greater than 2 times the ULN
* serum creatinine levels or more than 2mg/dL
* The patient requires current treatment for HIV with protease inhibitors.
* The patient is taking medication for a clinical diagnosis of gastrointestinal ulceration or has experienced melena or hematoemesis in the previous 3 weeks.
* The patient is a woman who is pregnant or lactating.
* The patient has received treatment with an investigation drug within 4 weeks of the planned 1st day of study treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2005-06; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Physicians Static Global (PSGA) Score | 87 Days
  The primary objective of the study is to evaluate the efficacy of oral escalating dosages of CEP-701 at 20, 40, 60, and 80 mg given twice daily (bid) in achieving complete or nearly clearing of psoriasis in patients with severe, recalcitrant, plaque-type psoriasis, as assessed by the Physicians Static Global (PSGA) at baseline and at the end of treatment. A PSGA score of 0 is defined as no evidence of plaque elevation, no evidence of erythema, and no evidence of scaling. A PSGA score of 5 is defined as plaque elevation (2.5 mm or greater)dusky to deep red coloration, very thick tenacious scale predominates.

SECONDARY OUTCOMES:
PSGA Change from Baseline | 87 days
  Change from baseline to the end of treatment (ie, day 85±2 PSGA measured on a scale of 0 to 5 at the end of treatment severity of itch measured on a severity scale of 0 to 5 at the 85±2 days) 0 meaning No itching - 5 Severe; constant itching; distressing; frequent disturbance of sleep; interferes with activities
Psoriasis Area and Severity Index (PASI) | 87 Days
  Psoriasis Area and Severity Index (PASI) 0=no involvement
  1=<10% involvement 2=10% to <30% involvement 3=30% to <50% involvement 4=50% to <70% involvement 5=70% to <90% involvement 6=90% to 100% involvement

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Wake Forest University, Winston-Salem, North Carolina
  - Texas Dermatology Rsch Inst, Dallas, Texas
  - Viginia Clinical Research, Norfolk, Virginia